CLINICAL TRIAL: NCT01459848
Title: A Randomized Controlled Trial of Block Play vs Dvd Viewing
Brief Title: Baby Dvd Effects on Cortisol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Dimitri Christakis, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Baby DVD study; Endowment (Other Grant/Funding Number: Adkins endowment)
Record Dates: First submitted 2011-10-20; First posted 2011-10-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Infant Development
Keywords: Salivary cortisol measured after DVD watching or block play

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- block play (Active Comparator): 30 minutes of block play with parent
  Interventions: Behavioral: block play
- baby dvd (Experimental): watch baby dvd with parent
  Interventions: Behavioral: baby dvd

INTERVENTIONS:
Behavioral: block play — 30 minutes of block play
  Arms: block play
Behavioral: baby dvd — 30 minutes of dvd viewing
  Arms: baby dvd

SUMMARY:
The investigators will do an experiment where 9-12 month old infants are randomized to 30 minutes of block play or 30 minutes of watching a baby DVD.

ELIGIBILITY:
Inclusion Criteria:

* 9-12 months of age

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
salivary cortisol | Baseline
  Study will be assessing babies' neuroendocrine responses to play vs TV viewing. Salivary cortisol, as an indicator of neuroendocrine response, will be measured over time with the intervals as specified under time frame. For each time point, investigator will adjust for prior ones in a repeated measures analysis.
salivary cortisol | 10 minutes post baseline
  Study will be assessing babies' neuroendocrine responses to play vs TV viewing. Salivary cortisol, as an indicator of neuroendocrine response, will be measured over time with the intervals as specified under time frame. For each time point, investigator will adjust for prior ones in a repeated measures analysis
salivary cortisol | 20 minutes post baseline
  Study will be assessing babies' neuroendocrine responses to play vs TV viewing. Salivary cortisol, as an indicator of neuroendocrine response, will be measured over time with the intervals as specified under time frame. For each time point, investigator will adjust for prior ones in a repeated measures analysis
salivary cortisol | 30 minutes post baseline
  Study will be assessing babies' neuroendocrine responses to play vs TV viewing. Salivary cortisol, as an indicator of neuroendocrine response, will be measured over time with the intervals as specified under time frame. For each time point, investigator will adjust for prior ones in a repeated measures analysis
salivary cortisol | 40 minutes post baseline
  Study will be assessing babies' neuroendocrine responses to play vs TV viewing. Salivary cortisol, as an indicator of neuroendocrine response, will be measured over time with the intervals as specified under time frame. For each time point, investigator will adjust for prior ones in a repeated measures analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Christakis, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle CHildrens Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Christakis DA, Liekweg K, Garrison MM, Wright JA. Infant video viewing and salivary cortisol responses: a randomized experiment. J Pediatr. 2013 May;162(5):1035-40. doi: 10.1016/j.jpeds.2012.10.032. Epub 2012 Nov 16. PMID 23164310